CLINICAL TRIAL: NCT00653068
Title: Treatment of Atypical Teratoid/Rhabdoid Tumors (AT/RT) of the Central Nervous System With Surgery, Intensive Chemotherapy, and 3-D Conformal Radiation
Brief Title: Combination Chemotherapy, Radiation Therapy, and an Autologous Peripheral Blood Stem Cell Transplant in Treating Young Patients With Atypical Teratoid/Rhabdoid Tumor of the Central Nervous System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0333; NCI-2009-00337 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000592812; 09-0058; COG-ACNS0333; ACNS0333 (Other: Children's Oncology Group); ACNS0333 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor
MeSH Terms: conditions — Rhabdoid Tumor | interventions — Radiotherapy, Conformal; Stem Cell Transplantation; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Methotrexate; merphos; Thiotepa; Vincristine

ARMS (2):
- Arm I (chemotherapy, autologous PBSC, 3D-CRT) (Experimental): Patients receive vincristine IV on days 1, 8, and 15; high-dose methotrexate IV on day 1; leucovorin calcium orally or IV; etoposide IV on days 4, 5, and 6; cyclophosphamide IV on days 4 and 5; cisplatin IV on day 6, and G-CSF IV or SC on day 7 until ANC recovers.
  Within 2-6 weeks after induction therapy or radiation therapy, patients receive high-dose carboplatin IV and high-dose thiotepa IV on days 1 and 2 and undergo autologous PBSC rescue on approximately day 4. Patients also receive G-CSF IV or SC once daily until ANC recovers. Treatment with consolidation therapy followed by stem cell rescue repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. After consolidation therapy, patients undergo 3D-CRT to the brain (and the spine if needed) 5 days a week for 5-6 weeks.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Thiotepa; Drug: Vincristine Sulfate
- Arm II (chemotherapy, 3D-CRT, autologous PBSC) (Experimental): Patients receive vincristine IV on days 1, 8, and 15; high-dose methotrexate IV on day 1; leucovorin calcium orally or IV; etoposide IV on days 4, 5, and 6; cyclophosphamide IV on days 4 and 5; cisplatin IV on day 6, and G-CSF IV or SC on day 7 until ANC recovers.
  Patients undergo 3D-CRT to the brain (and the spine if needed) 5 days a week for 5-6 weeks. Within 2-6 weeks after completion of radiation therapy, patients receive high-dose carboplatin IV and high-dose thiotepa IV on days 1 and 2 and undergo autologous PBSC rescue on approximately day 4. Patients also receive G-CSF IV or SC once daily until ANC recovers. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Thiotepa; Drug: Vincristine Sulfate

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSC rescue
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16
Biological: Filgrastim — Given IV or SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV or PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; Folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies the side effects of combination chemotherapy, 3-dimensional conformal radiation therapy, and an autologous peripheral blood stem cell transplant, and to see how well they work in treating young patients with atypical teratoid/rhabdoid tumor of the central nervous system. Giving high-dose chemotherapy before an autologous peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy or radiation therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 6-, 12-, and 24-month event-free survival and overall survival of children (birth to 21 years of age) with atypical teratoid/rhabdoid CNS tumors (AT/RT), diagnosed based on histology, immunophenotyping, and modern molecular and immunohistochemical analysis of INI1, treated with surgery, intensive chemotherapy combined with stem cell rescue, and radiation therapy.

II. To compare the outcome of very young patients (under 3 years old) on this study whose histologic diagnosis is AT/RT with infants identified as having AT/RT on POG-9233 and CCG-9921.

SECONDARY OBJECTIVES:

I. To determine the feasibility and toxicity of the proposed chemotherapy regimen in combination with radiation therapy.

II. To contribute tumor samples from which biologic and gene expression data can be developed to yield prognostic indicators and provide direction for future treatment strategies.

III. To develop a clinical and biologic database on which future studies can be based.

OUTLINE:

INDUCTION THERAPY AND STEM CELL HARVEST: Patients receive vincristine IV on days 1, 8, and 15 and high-dose methotrexate IV over 4 hours on day 1. Beginning 24 hours after the start of methotrexate, patients receive leucovorin calcium orally (PO) or IV every 6 hours until the serum methotrexate level is < 0.1 micromoles. Patients then receive etoposide IV over 1 hour on approximately days 4, 5, and 6, cyclophosphamide IV over 1 hour on approximately days 4 and 5, and cisplatin IV over 6 hours on approximately day 6*. Patients also receive filgrastim (G-CSF) IV or subcutaneously (SC) once daily beginning on day 7 and continuing until ANC recovers. When ANC is > 1,000/uL post nadir, patients receive G-CSF twice daily for stem cell mobilization. Approximately 2-4 days, later peripheral blood stem cells are harvested once daily, as needed, after each course of induction therapy until a total of 6 x 10^6 CD34+ cells/kg have been collected. Treatment repeats every 21 days for 2 courses.

After completion of induction therapy, patients are re-evaluated. Patients with progressive disease are removed from study. Patients with radiographic evidence of residual tumor are encouraged to undergo second-look surgery prior to proceeding to radiotherapy or consolidation therapy; patients with complete response, partial response, or stable disease are assigned to 1 of 2 arm.

ARM I ((patients less than 6 months, infratentorial site with M0 involvement or patients less than 12 months, supratentorial site with M0 involvement or patients with disseminated disease of any primary site or age):

CONSOLIDATION THERAPY AND STEM CELL RESCUE: Within 2-6 weeks after completion of induction therapy, patients begin consolidation therapy. Patients receive high-dose carboplatin IV over 4 hours and high-dose thiotepa IV over 2 hours on days 1 and 2 and undergo autologous peripheral blood stem cell (PBSC) rescue on approximately day 4. Patients also receive G-CSF IV or SC once daily beginning 24 hours after stem cell infusion and continuing until ANC recovers. Treatment with consolidation therapy followed by stem cell rescue repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

RADIATION THERAPY: Patients undergo 3-dimensional conformal radiotherapy (3D-CRT) to the brain (and the spine if needed) 5 days a week for 5-6 weeks.

ARM II (patients greater than or equal to 6 months, infratentorial site with M0 involvement or patients greater than or equal to 12 months, supratentorial site with M0 involvement): Patients undergo 3D-CRT as in Arm I. Within 2-6 weeks after completion of radiation therapy, patients receive consolidation therapy and stem cell rescue as in Arm I

NOTE: *The administration of etoposide, cyclophosphamide, and cisplatin are dependant on the prior clearance of methotrexate to a level of < 0.1 micromoles.

After completion of study treatment, patients are followed periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CNS atypical teratoid/rhabdoid tumor (AT/RT) or tumors that have a mutation of the INI1 gene (even if the tumor does not have the usual histologic characteristics of AT/RT)

  * Patients with extra neural metastasis (M4) or renal rhabdoid tumors are not eligible
  * Patients with MRI evidence of spinal disease are eligible
* Must have undergone definitive surgery in the past 31 days
* Cranial MRI (with and without gadolinium) must be done pre-operatively

  * Post-operatively, cranial MRI (with and without gadolinium) must be done, preferably within 48 hours of surgery or 10-28 days after surgery
* Entire spinal MRI must be obtained either pre-operatively (with gadolinium) or post-operatively (10-28 days after surgery), prior to study enrollment (with and without gadolinium)
* Life expectancy > 8 weeks
* ANC > 1,000/uL
* Platelet count > 100,000/uL (transfusion independent)
* Hemoglobin > 8 g/dL (RBC transfusions allowed)
* Creatinine clearance (minimum of 12-24 hour urine collection) or radioisotope GFR >= 60 mL/min
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* AST and ALT < 2 times ULN for age
* Shortening fraction of >= 27% by echocardiogram OR ejection fraction of >= 47% by radionuclide angiogram
* No evidence of dyspnea at rest
* Pulse oximetry > 94% on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior radiotherapy or chemotherapy except for the following:

  * Patients enrolled on protocol ACNS0334 whose tumors demonstrate the INI1 gene mutation are eligible to transfer to this study even if they have received one course of induction therapy (these patients must be re-consented to treatment and restaged)
  * Prior corticosteroids allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02-10 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa T Reddy, Principal Investigator — Children's Oncology Group
Locations (94):
- United States (87):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Mazzarella J, Heathcock JC. A Randomized Feasibility Study of Rehabilitation Targeting Upper Extremity Function and Participation Using Hippotherapy and the Equine Environment for Children with Cerebral Palsy and Autism Spectrum Disorder. J Integr Complement Med. 2025 Feb;31(2):196-208. doi: 10.1089/jicm.2024.0292. Epub 2024 Nov 8. PMID 39515374
- [Derived] Reddy AT, Krailo MD, Buxton AB, Strother DR, Huang A, Zhou T, Judkins AR, Burger PC, Pollack IF, Williams-Hughes C, Fouladi M, Ho B, Mazewski CM, Lewis VA, Vezina LG, Booth TN, Mahajan A. Reply to S.A. Upadhyaya. J Clin Oncol. 2020 Oct 1;38(28):3353-3354. doi: 10.1200/JCO.20.01573. Epub 2020 Jul 30. No abstract available. PMID 32730180
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Within 2-6 weeks after induction therapy or radiation therapy, patients receive high-dose carboplatin IV and high-dose thiotepa IV on days 1 and 2 and undergo autologous PBSC rescue on approximately day 4. Patients also receive G-CSF IV or SC once daily until ANC recovers.
  Consolidation therapy followed by stem cell rescue repeats every 28 days for 3 courses (C) and 3D-CRT to the brain (and the spine if needed) 5 days a week for 5-6 weeks (R), the order of which depends on patient age, in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment
Started | 70
Completed | 20
Not Completed | 50
Not completed — Death | 9
Not completed — Lack of Efficacy | 34
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Groups:
- Stratum I: Infants (<36 months of age) with tumor histology and immunohistochemical analysis diagnostic of AT/RT.
- Stratum II: Infants with INI1 mutation only based diagnosis (histology is not consistent with AT/RT).
- Stratum III: Older children (greater than 36 months of age) with tumor histology and immunohistochemical analysis diagnostic of AT/RT.
- Stratum IV: Older children with INI1 mutation only based diagnosis.
- Total: Total of all reporting groups
Arm/Group | Stratum I | Stratum II | Stratum III | Stratum IV | Total
Number analyzed (Participants) | 58 | 0 | 12 | 0 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58 |  | 12 |  | 70
  Between 18 and 65 years | 0 |  | 0 |  | 0
  >=65 years | 0 |  | 0 |  | 0
Age, Continuous [Median (Full Range); unit: years] | 1 [0 to 2] |  | 4 [3 to 14] |  | 1 [0 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 |  | 8 |  | 36
  Male | 30 |  | 4 |  | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 |  | 5 |  | 20
  Not Hispanic or Latino | 39 |  | 7 |  | 46
  Unknown or Not Reported | 4 |  | 0 |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  | 0 |  | 1
  Asian | 1 |  | 2 |  | 3
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 |  | 0
  Black or African American | 7 |  | 1 |  | 8
  White | 40 |  | 7 |  | 47
  More than one race | 0 |  | 0 |  | 0
  Unknown or Not Reported | 9 |  | 2 |  | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6 |  | 2 |  | 8
  United States | 51 |  | 10 |  | 61
  Australia | 1 |  | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Estimated 4-year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients without an event are censored at last contact.
Time Frame: Up to 4 years after study enrollment
Population: One patient was ineligible in stratum I and one patient was ineligible in stratum III. There were no patients enrolled in Stratum 2 or 4.
Measure: Number (95% Confidence Interval); unit: Estimated probability
Arm/Group | Stratum I | Stratum III
Number analyzed (Participants) | 57 | 11
Estimated probability | 0.3401 [0.2174 to 0.4666] | 0.4500 [0.1267 to 0.7345]

2. Primary Outcome: Overall Survival (OS)
Description: Estimated 4-year survival, where survival is calculated as the time from study enrollment to death from any cause or last follow-up alive whichever occurs first. Kaplan-Meier method is used for estimation. Patients alive at last contact are censored.
Time Frame: Up to 4 years after study enrollment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Estimated Probability
Arm/Group | Stratum I | Stratum III
Number analyzed (Participants) | 57 | 11
Estimated Probability | 0.3888 [0.2582 to 0.5173] | 0.5486 [0.1873 to 0.8064]

3. Primary Outcome: Toxic Death
Description: The number of patients who experience death that is considered to be primarily attributable to complications of treatment.
Time Frame: During and after completion of study treatment up to 1 year after enrollment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum I | Stratum III
Number analyzed (Participants) | 57 | 11
Participants | 3 | 1

4. Secondary Outcome: Non-hematological Toxicity Associated With Chemotherapy: Grade 3 or Higher During Protocol Therapy
Description: Number of Participants with Nonhematological Toxicity Associated With Chemotherapy: Grade 3 or Higher During Protocol Therapy.
Time Frame: During protocol therapy up to 1 year after enrollment.
Population: 68 eligible patients were evaluable
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Experimental
Arm/Group | All Patients
Number analyzed (Participants) | 68
Participants
  Acidosis | 1
  Acute kidney injury | 1
  Apnea | 2
  Adult respiratory distress syndrome | 1
  Aspiration | 3
  Atelectasis | 1
  Catheter related infection | 2
  Central nervous system necrosis | 1
  Dehydration | 1
  Diarrhea | 1
  Dissmeminated intravascular coagulation (DIC) | 1
  Enterocolitis | 1
  Febrile neutropenia | 6
  Hearing impairment | 1
  Hematuria | 1
  Hydrocephalus | 1
  Hypernatremia | 1
  Hypoalbuminemia | 1
  Hypocalcemia | 3
  Hypoglycemia | 2
  Hypokalemia | 9
  Hyponatremia | 2
  Hypophosphatemia | 2
  Hypotension | 4
  Hypoxia | 6
  Increased Alanine aminotransferase | 5
  Increased Aspartate aminotransferase | 4
  Increased Lipase | 1
  Intracranial hemorrhage | 2
  ntraoperative venous injury | 1
  Laryngospasm | 1
  Left ventricular systolic dysfunction | 1
  Lung infection | 3
  Multi-organ failure | 1
  Mucositis oral | 3
  Poisoning and procedural complications | 1
  Other gastrointestinal disorders | 1
  Other infection | 7
  Pneumonitis | 2
  Productive cough | 1
  Pulmonary edema | 1
  Recurrent laryngeal nerve palsy | 1
  Renal calculi | 1
  Respiratory failure | 3
  Seizure | 2
  Sepsis | 6
  Sinus tachycardia | 2
  Stridor | 2
  Upper respiratory infection | 1
  Vascular access complication | 1
  Voice alteration | 1
  Vomiting | 1
  Weight loss | 1

ADVERSE EVENTS:
Description: There were no patients enrolled in Stratum 2 or 4.
Arm/Group | Stratum I | Stratum III
Serious Adverse Events (participants affected / at risk) | 7/57 | 0/11
Other Adverse Events (participants affected / at risk) | 43/57 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum I (N=57) | Stratum III (N=11)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum I (N=57) | Stratum III (N=11)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 7 (7) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 18 (18) | 1 (1)
Neutrophil count decreased (Investigations) | 37 (37) | 5 (5)
Platelet count decreased (Investigations) | 31 (31) | 5 (5)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 30 (30) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.